CLINICAL TRIAL: NCT03049761
Title: Evaluation of the Safety of a Water Flosser on Gingival and Epithelial Tissue at Different Pressure Settings
Brief Title: Water Flosser vs String Floss vs Manual Toothbrush Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All Sum Research Center Ltd. (Other)
Collaborators: Water Pik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-WP-1
Record Dates: First submitted 2017-02-07; First posted 2017-02-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2017-02

CONDITIONS: Soft Tissue Injuries
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Intervention Model Description: This is a examiner-masked, 3-treatment, randomized clinical trial comparing the safety of different oral hygiene regimens.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Water Flosser (Active Comparator): Power interdental Cleaning Device
  Interventions: Device: Water Flosser
- String floss (Active Comparator): Manual interdental cleaning device
  Interventions: Device: String Floss
- Manual Toothbrush (Active Comparator): ADA standard manual toothbrush
  Interventions: Device: Manual Toothbrush

INTERVENTIONS:
Device: Water Flosser — Power interdental cleaner
  Arms: Water Flosser
Device: String Floss — Mechanical interdental cleaner
  Arms: String floss
Device: Manual Toothbrush — ADA standard soft bristle toothbrush
  Arms: Manual Toothbrush

SUMMARY:
Evaluation of the Safety of a Water Flosser on Gingival and Epithelial Tissue at Different Pressure Settings

DETAILED DESCRIPTION:
This study is designed to add to the safety data by measuring, Oral Soft tissue, Clinical Attachment Levels and Probing Pocket Depths on different pressure settings at different time points over a 6 week period. Data will be collected at Baseline, 2 week, 4 week and 6 week time frames.

ELIGIBILITY:
Inclusion Criteria:

* Written consent prior to participation
* Good general health and non smoker
* Have scorable Ramfjord's teeth

Exclusion Criteria:

* Probing depth >4mm on Ramfjord's teeth
* Moderate to severe gingivitis
* Advanced periodontitis
* Medications that impact soft tissue.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Levels | 6 weeks
  Measurement from the junction Epithelium to the cemento enamel junction

SECONDARY OUTCOMES:
Probing pocket depth | 6 weeks
  Measurement from the junction Epithelium to the free gingival margin

IPD SHARING:
Plan to Share IPD: No